CLINICAL TRIAL: NCT03032614
Title: Phase II Clinical Trial on the Combination of Carboplatin, Eribulin and Veliparib in Stage IV Cancer Patients With Homologous Recombination Deficiency
Brief Title: Combination of Carboplatin, Eribulin and Veliparib in Stage IV Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Virginia G. Kaklamani, Clinical Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS#16-0133; 17-166H (Other: UTHSCSA)
Record Dates: First submitted 2017-01-23; First posted 2017-01-26 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer Stage IV; Ovarian Cancer; BRCA1 Mutation; BRCA2 Mutation
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; eribulin; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of Carboplatin, Eribulin, and Veliparib (Experimental): Eribulin will be administered intravenously (IV) on days 1 and 8 of each cycle at a dose of 1.1 mg/m2 over a 2-5 minute time period; on cycle day 1. Carboplatin will be administered intravenously at a dose of AUC 5 on day 1 of each cycle, over 30 min, immediately following eribulin infusion, per institutional guidelines. Veliparib will be given at 120 mg bid (two times a day), on days 2-12 for the first cycle of the safety run-in period and thereafter at 240 mg bid.
  Interventions: Drug: Carboplatin; Drug: Eribulin; Drug: Veliparib

INTERVENTIONS:
Drug: Carboplatin — Carboplatin is a second generation tetravalent organic platinum compound. Similar to cisplatin, carboplatin produces predominantly interstrand DNA crosslinks as opposed to DNA-protein crosslinks. Carboplatin is cell-cycle non-specific.
  Other Names: Paraplatin
Drug: Eribulin — Eribulin Mesylate is a synthetic halichondrin analog.
  Other Names: Halaven; E7389
Drug: Veliparib — Veliparib is a potent PARP inhibitor that delays the repair of DNA damage induced by chemotherapeutics.
  Other Names: ABT-888

SUMMARY:
This is a phase II clinical trial of the combination of carboplatin, eribulin, and Veliparib.

DETAILED DESCRIPTION:
This is a Phase II, non-randomized, open-label, Clinical Trial on the Combination of Carboplatin, Eribulin, and Veliparib in Patients with BRCA-related Cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have archival biopsy specimens (preferably from metastatic disease) available for research tests. If a suitable biopsy specimen is not available, patients will be asked to undergo a research biopsy to procure tissue
* Patients must be >/= 18 years
* Females of childbearing potential must not have had unprotected sexual intercourse within 30 days prior to study entry and must agree to use a highly effective method of contraception. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation
* Patients must have an ECOG performance status 0-1
* Patients may have had a prior diagnosis of cancer if it has been > 5 years since their last treatment for that cancer
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes ≥ 3,000/uL
  * Absolute neutrophil count ≥ 1,500/uL
  * Platelets ≥ 100,000/uL
  * Creatinine within normal limits or creatinine clearance ≥30
* Patients must be able to swallow and retain oral medication
* Patients who were receiving prior systemic therapy: Prior treatment related side effects must have resolved to < Grade 2 severity (except alopecia and infertility)
* All patients must have given signed, informed consent prior to registration on study
* Patients must have stage IV breast or stage III and IV ovarian cancer (including platinum sensitive disease)
* Patients must have BRCA1/2 deleterious mutations, PTEN deficiency, or cancer with a high HRD score as assessed by Myriad's assay
* Patients must have measurable disease per RECIST 1.1 criteria (see above for definition)
* Patients may not have received more than 3 chemotherapeutic regimens for metastatic disease
* Patients may not have received treatment with prior carboplatin, eribulin or a PARP inhibitor

Exclusion Criteria:

* Women who are pregnant or lactating are not eligible
* Patients who are undergoing concomitant radiotherapy are not eligible
* Patients who are receiving any other investigational agents or concurrent anticancer therapy are not eligible
* Previous systemic treatment is allowed with a 21 day washout period prior to registration
* Patients who are taking any herbal (alternative) medicines are not eligible. Patients must be off any such medications by the time of registration
* Patients with known brain metastases are not eligible for participation unless the following are met:

  * Brain metastases are treated (either with surgical excision, stereotactic radiosurgery or radiotherapy and have been stable for at least 4 weeks (MRI documented)
  * Patient is asymptomatic and has discontinued corticosteroids if taken for that purpose
* Patients with any of the following conditions or complications are NOT eligible for participation:

  * GI tract disease resulting in an inability to take oral medication
  * Malabsorption syndrome
  * Require IV alimentation
  * History of prior surgical procedures affecting absorption
  * Uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
  * Hypersensitivity of any of the components of Veliparib, carboplatin, eribulin
  * History of significant neurological (no neuropathy > Grade 2) or psychiatric disorders.
  * Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).
  * Significant non-neoplastic renal disease.
  * Immunocompromised subjects, including subjects known to be infected with human immunodeficiency virus (HIV).
  * Uncontrolled endocrine diseases (e.g., diabetes mellitus, hypothyroidism or hyperthyroidism, adrenal disorder) i.e., requiring relevant changes in medication within the last month or hospital admission within the last three months
  * Active infection requiring systemic therapy.
  * Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment.
  * Prolongation of QTc interval to > 480 msec when electrolytes balance is normal.
  * Major surgery within 4 weeks prior to the first dose of study drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must have breast and ovarian cancer
Enrollment: 0 (Actual)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature and severity of adverse events and serious adverse events, graded according to NCI - Common Toxicity Criteria for Adverse Events version (4.03) | Approximately 1.5 years
  Graded according to NCI - Common Toxicity Criteria for Adverse Events version (4.03)
Tumor response assessed using RECIST 1.1 guidelines | Measured every 6 weeks for 21 day cycles for the duration of study treatment, estimated to be less than one year
  Response will be assessed in this study via physical exam and imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kaklamani, MD, Principal Investigator — UT Health San Antonio

IPD SHARING:
Plan to Share IPD: Undecided